CLINICAL TRIAL: NCT00350779
Title: A Phase III Randomized, Placebo-Controlled Clinical Trial to Study the Safety and Efficacy of the Addition of Sitagliptin (MK0431) in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Combination Therapy With Metformin and a PPARg Agonist
Brief Title: Sitagliptin Metformin/PPARg Agonist Combination Therapy Add-on (0431-052)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-052; MK0431-052; 2006_507
Record Dates: First submitted 2006-07-07; First posted 2006-07-11 (Estimated); Results first posted 2009-07-03 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Rosiglitazone; Metformin; Glipizide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Sitagliptin
  Interventions: Drug: sitagliptin; Drug: rosiglitazone; Drug: metformin; Drug: glipizide
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo; Drug: rosiglitazone; Drug: metformin; Drug: glipizide

INTERVENTIONS:
Drug: sitagliptin — Sitagliptin 100mg tablet each day for 54 weeks. All subjects will be given placebo to sitagliptin for a 2 week period.
  Other Names: Januvia
  Arms: 1
Drug: Comparator: Placebo — Placebo to sitagliptin 100mg tablet each day for 54 weeks.
  Arms: 2
Drug: rosiglitazone — Subjects taking 4mg or greater rosiglitazone at screening will enter a 6 week stable dose period followed by a 54 week treatment period. Subjects who are taking less than 4mg/day or no rosiglitazone at screening will be titrated to a stable dose of at least 4mg over a a maximum of 8 weeks followed by a dose stable period of up to 12 weeks then a 54 week treatment period. Total treatment will be up to 77 weeks.
  Other Names: Avandia
Drug: metformin — Subjects taking 1500mg or greater metformin at screening will enter a 6 week stable dose period followed by a 54 week treatment period. Subjects who are taking less than 1500mg/day or no metformin at screening will be titrated to a stable dose of at least 1500mg over a a maximum of 8 weeks followed by a dose stable period of up to 12 weeks then a 54 week treatment period. Total treatment will be up to 77 weeks.
Drug: glipizide — Subjects not meeting specific glycemic controls during the 54-week treatment period will use glipizide as rescue therapy. Glipizide will be titrated in 5mg doses up to a maximum 40mg each day. (In Canada, the rescue therapy will be a sulfonylurea agent marketed in that country.)
  Other Names: Glucotrol

SUMMARY:
A clinical study to determine the safety and efficacy of sitagliptin in patients with Type 2 Diabetes Mellitus who have inadequate glycemic control on metformin/peroxisome proliferator-activated receptor gamma (PPARg) agonist combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient has type 2 diabetes mellitus
* Patient is inadequately controlled while taking two oral antidiabetic medications

Exclusion Criteria:

* Patient has a history of type 1 diabetes mellitus or history of ketoacidosis
* Patient required insulin therapy within the prior 3 months
* Patient has been taking Byetta (R) (exenatide) within the prior 3 months

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2006-06-12 (Actual); Primary Completion 2007-09-25 (Actual); Study Completion 2008-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Dobs AS, Goldstein BJ, Aschner P, Horton ES, Umpierrez GE, Duran L, Hill JS, Chen Y, Golm GT, Langdon RB, Williams-Herman DE, Kaufman KD, Amatruda JM, Ferreira JC. Efficacy and safety of sitagliptin added to ongoing metformin and rosiglitazone combination therapy in a randomized placebo-controlled 54-week trial in patients with type 2 diabetes. J Diabetes. 2013 Mar;5(1):68-79. doi: 10.1111/j.1753-0407.2012.00223.x. PMID 22742523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III
  First Patient In: 29-Aug-06. Last Patient Enrolled: 23-Mar-07. Last Patient Last Visit: 27-May-08; 41 study centers worldwide
Pre-assignment Details: Patients 18-78 years of age with T2DM and inadequate glycemic control (HbA1c ≥7.5 and ≤11.0%) who were on stable doses of rosiglitazone (≥4 mg/day) and metformin (≥1500 mg/day) after an up to 20-week dose-titration and stabilization period were eligible to enter the 54-week study.
Groups:
- Sitagliptin 100 mg: The Sitagliptin 100 mg group includes data from patients randomized to receive treatment with 100 mg oral tablets of sitagliptin once daily (blinded) in addition to ongoing treatment with open-label rosiglitazone 4 mg oral tablets (4 to 8 mg/day) and open-label metformin 500 mg oral tablets (≥1500 mg/day).
- Placebo: The Placebo group includes data from patients randomized to receive treatment with placebo to sitagliptin 100 mg tablet once daily (blinded) in addition to ongoing treatment with open-label rosiglitazone 4 mg oral tablets (4 to 8 mg/day) and open-label metformin 500 mg oral tablets (≥1500 mg/day).
Period: Overall Study
Arm/Group | Sitagliptin 100 mg | Placebo
Started | 170 | 92
Completed | 148 | 71
Not Completed | 22 | 21
Not completed — Adverse Event | 4 | 2
Not completed — Lack of Efficacy | 0 | 4
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 2 | 4
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 9 | 8
Not completed — Patient Moved | 2 | 1
Not completed — Non-compliance with study procedures | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 100 mg | Placebo | Total
Number analyzed (Participants) | 170 | 92 | 262
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (8.8) | 54.8 (9.5) | 54.5 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 37 | 111
  Male | 96 | 55 | 151
Race/Ethnicity [Number; unit: participants]
  White | 82 | 51 | 133
  Black | 7 | 3 | 10
  Hispanic | 13 | 10 | 23
  Asian | 58 | 24 | 82
  Other | 10 | 4 | 14
HbA1c (Hemoglobin A1c) [Mean (Standard Deviation); unit: Percent] | 8.8 (1.0) | 8.7 (1.0) | 8.8 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Hemoglobin A1C) at Week 18
Description: HbA1c is measured as a percent. Thus, this change from baseline reflects the Week 18 HbA1c percent minus the Week 0 HbA1c percent.
Time Frame: Baseline and 18 Weeks
Population: The Full Analysis Set (FAS) included all patients with a baseline value and ≥1 post-baseline value for this outcome. Data following glycemic rescue were treated as missing. For FAS patients with no data at Week 18, the last non-baseline observed measurement was carried forward to Week 18.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 168 | 88
Percent | -1.03 [-1.17 to -0.90] | -0.31 [-0.50 to -0.13]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment; baseline; prior anti-hyperglycemic therapy; Mean Difference (Net) = -0.72, 95% CI [-0.95 to -0.49], Standard Deviation 0.87

2. Secondary Outcome: Change From Baseline in FPG (Fasting Plasma Glucose) at Week 18
Description: Change from baseline at Week 18 is defined as Week 18 minus Week 0
Time Frame: Baseline and 18 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 169 | 89
mg/dL | -30.7 [-35.5 to -26.0] | -11.7 [-18.3 to -5.1]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment; baseline; prior anti-hyperglycemic therapy; Mean Difference (Net) = -19.0, 95% CI [-27.2 to -10.9], Standard Deviation 31.3

3. Secondary Outcome: Change From Baseline in 2-hour PMG (Post-meal Glucose) at Week 18
Description: Change from baseline at Week 18 is defined as Week 18 minus Week 0
Time Frame: Baseline and Week 18
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 142 | 75
mg/dL | -59.9 [-67.1 to -52.6] | -22.0 [-32.1 to -12.0]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment; baseline; prior anti-hyperglycemic therapy; Mean Difference (Net) = -37.9, 95% CI [-50.2 to -25.5], Standard Deviation 43.7

4. Secondary Outcome: Change From Baseline in HbA1c (Hemoglobin A1C) at Week 54
Description: HbA1c is measured as a percent. Thus, this change from baseline reflects the Week 54 HbA1c percent minus the Week 0 HbA1c percent.
Time Frame: Baseline and Week 54
Population: The Full Analysis Set (FAS) included all patients with a baseline value and ≥1 post-baseline value for this outcome. Data following glycemic rescue were treated as missing. For FAS patients with no data at Week 54, the last non-baseline observed measurement was carried forward to Week 54.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 168 | 88
Percent | -1.05 [-1.21 to -0.89] | -0.28 [-0.50 to -0.05]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment; baseline; prior anti-hyperglycemic therapy; Mean Difference (Net) = -0.77, 95% CI [-1.04 to -0.50], Standard Deviation 1.04

5. Secondary Outcome: Change From Baseline in FPG (Fasting Plasma Glucose) at Week 54
Description: Change from baseline at Week 54 is defined as Week 54 minus Week 0
Time Frame: Baseline and Week 54
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 169 | 89
mg/dL | -28.0 [-33.3 to -22.8] | -10.7 [-18.0 to -3.3]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment; baseline; prior anti-hyperglycemic therapy; Mean Difference (Net) = -17.4, 95% CI [-26.4 to -8.4], Standard Deviation 34.6

6. Secondary Outcome: Change From Baseline in 2-hour PMG (Post-meal Glucose) at Week 54
Description: Change from baseline at Week 54 is defined as Week 54 minus Week 0.
Time Frame: Baseline and Week 54
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 147 | 77
mg/dL | -50.7 [-59.1 to -42.4] | -16.6 [-28.2 to -5.0]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment; baseline; prior anti-hyperglycemic therapy; Mean Difference (Net) = -34.1, 95% CI [-48.4 to -19.9], Standard Deviation 51.0

ADVERSE EVENTS:
Groups:
- Sitagliptin 100 mg Data Through Week 18: The Sitagliptin 100 mg group includes data from patients randomized to receive treatment with 100 mg oral tablets of sitagliptin once daily (blinded) in addition to ongoing treatment with open-label rosiglitazone 4 mg oral tablets (4 to 8 mg/day) and open-label metformin 500 mg oral tablets (≥1500 mg/day).
- Placebo Data Through Week 18: The Placebo group includes data from patients randomized to receive treatment with placebo to sitagliptin 100 mg tablet once daily (blinded) in addition to ongoing treatment with open-label rosiglitazone 4 mg oral tablets (4 to 8 mg/day) and open-label metformin 500 mg oral tablets (≥1500 mg/day).
Arm/Group | Sitagliptin 100 mg Data Through Week 18 | Placebo Data Through Week 18 | Sitagliptin 100 mg Data Through Week 54 | Placebo Data Through Week 54
Serious Adverse Events (participants affected / at risk) | 2 | 2 | 14 | 4
Other Adverse Events (participants affected / at risk) | 20 | 14 | 70 | 35
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Sitagliptin 100 mg Data Through Week 18 | Placebo Data Through Week 18 | Sitagliptin 100 mg Data Through Week 54 | Placebo Data Through Week 54
Any Cardiac Disorders (Cardiac disorders) | 0/170 | 0/92 | 2/170 | 0/92
Myocardial Infarction (Cardiac disorders) | 0/170 | 0/92 | 2/170 | 0/92
Any Ear And Labyrinth Disorders (Ear and labyrinth disorders) | 0/170 | 0/92 | 1/170 | 0/92
Vertigo (Ear and labyrinth disorders) | 0/170 | 0/92 | 1/170 | 0/92
Any Hepatobiliary Disorders (Hepatobiliary disorders) | 0/170 | 0/92 | 1/170 | 0/92
Biliary Colic (Hepatobiliary disorders) | 0/170 | 0/92 | 1/170 | 0/92
Any Infections And Infestations (Infections and infestations) | 0/170 | 0/92 | 1/170 | 0/92
Urinary Tract Infection (Infections and infestations) | 0/170 | 0/92 | 1/170 | 0/92
Any Injury, Poisoning And Procedural Complications (Injury, poisoning and procedural complications) | 0/170 | 0/92 | 0/170 | 1/92
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0/170 | 0/92 | 0/170 | 1/92
Any Musculoskeletal And Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 1/170 | 0/92 | 3/170 | 0/92
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1/170 | 0/92 | 2/170 | 0/92
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0/170 | 0/92 | 1/170 | 0/92
Any Neoplasms Benign, Malignant And Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/170 | 1/92 | 4/170 | 2/92
Astrocytoma Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/170 | 0/92 | 0/170 | 1/92
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/170 | 1/92 | 1/170 | 1/92
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/170 | 0/92 | 1/170 | 0/92
Neurilemmoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/170 | 0/92 | 1/170 | 0/92
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/170 | 0/92 | 1/170 | 0/92
Any Nervous System Disorders (Nervous system disorders) | 0/170 | 0/92 | 2/170 | 0/92
Cerebrovascular Accident (Nervous system disorders) | 0/170 | 0/92 | 1/170 | 0/92
Diabetic Neuropathy (Nervous system disorders) | 0/170 | 0/92 | 1/170 | 0/92
Any Psychiatric Disorders (Psychiatric disorders) | 0/170 | 1/92 | 0/170 | 1/92
Suicidal Ideation (Psychiatric disorders) | 0/170 | 1/92 | 0/170 | 1/92
Any Renal And Urinary Disorders (Renal and urinary disorders) | 0/170 | 0/92 | 1/170 | 0/92
Renal Colic (Renal and urinary disorders) | 0/170 | 0/92 | 1/170 | 0/92
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Sitagliptin 100 mg Data Through Week 18 | Placebo Data Through Week 18 | Sitagliptin 100 mg Data Through Week 54 | Placebo Data Through Week 54
Any Gastrointestinal Disorders (Gastrointestinal disorders) | 0/170 | 0/92 | 8/170 | 5/92
Diarrhoea (Gastrointestinal disorders) | 0/170 | 0/92 | 8/170 | 5/92
Any General Disorders And Administration Site Conditions (General disorders) | 0/170 | 0/92 | 15/170 | 5/92
Oedema Peripheral (General disorders) | 0/170 | 0/92 | 15/170 | 5/92
Any Infections And Infestations (Infections and infestations) | 20/170 | 10/92 | 46/170 | 15/92
Nasopharyngitis (Infections and infestations) | 10/170 | 4/92 | 18/170 | 9/92
Upper Respiratory Tract Infection (Infections and infestations) | 10/170 | 6/92 | 28/170 | 6/92
Any Musculoskeletal And Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 0/170 | 5/92 | 7/170 | 5/92
Back Pain (Musculoskeletal and connective tissue disorders) | 0/170 | 5/92 | 7/170 | 5/92
Any Nervous System Disorders (Nervous system disorders) | 0/170 | 0/92 | 14/170 | 8/92
Dizziness (Nervous system disorders) | 0/170 | 0/92 | 6/170 | 5/92
Headache (Nervous system disorders) | 0/170 | 0/92 | 10/170 | 4/92
Any Respiratory, Thoracic And Mediastinal Disorders (Nervous system disorders) | 0/170 | 0/92 | 7/170 | 7/92
Cough (Respiratory, thoracic and mediastinal disorders) | 0/170 | 0/92 | 7/170 | 7/92

LIMITATIONS AND CAVEATS:
Non-serious adverse event results represent those events included in the primary safety analysis for this study (events occurred prior to initiation of glycemic rescue therapy). Site 0520039 was non-compliant with GDP, data was removed from analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.